CLINICAL TRIAL: NCT05175716
Title: Organizational Impact of Rapid Screening for COVID-19 by Delocalized Biology in the Birth Room
Acronym: DELOCOVIDMATER
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: DELOCOVIDMATER
Record Dates: First submitted 2021-12-31; First posted 2022-01-04 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-06

CONDITIONS: COVID-19; Labor
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
COVID-19 disease, caused by SARS-CoV-2 first appeared in China, and then spread worldwide. In December 2019, a group of patients with pneumonia of unknown origin were infected after exposure to the market in Wuhan, Hubei Province, China. Very quickly, a new coronavirus was isolated from a sample of a patient's lower respiratory tract and the complete genome of the virus was sequenced. This new coronavirus, named Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) for its genetic homology with SARS-CoV, showed a global extension. Thus, on January 30, 2020, the World Health Organization (WHO) announced the outbreak of COVID-19 as an international public health threat, and then in March 2020, the global situation escalated to a pandemic. Johns Hopkins University reported over 7,600,000 cases of infection and over 427,000 deaths as of June 13, 2020. Due to the rapid progression of the COVID-19 pandemic and the limited molecular testing capabilities at the laboratory level, the concept of molecular testing for off-site biology examination appears relevant. Indeed, the urgent need for increased testing for COVID-19 has been clearly identified as an essential element of the strategy to combat the coronavirus worldwide. Indeed, COVID-19 represents a major public health problem currently causing rapidly increasing numbers of infections and significant morbidity and mortality worldwide. As of September 3, 2021, more than 200 million people worldwide have been infected with SARS-CoV-2 and more than 4.5 million have died according to data collected by Johns Hopkins University. Early detection with a sensitive COVID-19 technique is essential to ensure rapid and appropriate patient management, contain the epidemic, and better understand the global epidemiology of the virus. To date, laboratory diagnostics have relied primarily on amplification and detection of viral gene sequences in upper respiratory tract specimens performed in a centralized laboratory. A new test (ID NOW COVID-19) is based on isothermal amplification at 56°C of the gene encoding the RdRp RNA polymerase. This molecular biology test can be performed as an off-site medical examination (EBMD), providing a result in less than 13 minutes directly in the clinical department. This rapidity could allow a more rapid management, isolation and "filiarization" of COVID-19 patients.

To our knowledge, there is no study available in the literature evaluating the impact of a rapid examination in delocalized biology on the organization of the management of pregnant women in the delivery room. The objective of this work is to evaluate the organizational impact of parturients who have received a rapid test for SARS-CoV-2.

The primary objective is to evaluate the impact of the use of the ID NOW COVID-19 test on the length of stay of parturients in the delivery room.

The secondary objectives are to evaluate the time to result, time to isolation and user satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Parturient whose age is ≥ 18 years
* Parturient in spontaneous labor
* French speaking parturient

Exclusion Criteria:

* Parturient under guardianship or curatorship
* Parturient deprived of liberty
* Parturient under court protection
* Parturient objecting to the use of her data for this research

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parturient whose age is ≥ 18 years, in spontaneous labor betwenn July 2020 and July 2021.
Sampling Method: Non-Probability Sample
Enrollment: 2447 (Actual)
Dates: Start 2022-01-14 (Actual); Primary Completion 2022-08-14 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Impact of the use of the ID NOW COVID-19 test on the length of stay of parturients in the delivery room | Day 1
  This outcome corresponds to the time of presence of the parturient in the birth room.

SECONDARY OUTCOMES:
Rendering time of the result | Day 1
  This outcome corresponds to the rendering time of the result.
Time to implement isolation | Day 1
  This outcome corresponds to the time to implement isolation.
User satisfaction | Day 1
  This outcome corresponds to the user satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude NGUYEN VAN, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France

REFERENCES:
- [Background] Zhu N, Zhang D, Wang W, Li X, Yang B, Song J, Zhao X, Huang B, Shi W, Lu R, Niu P, Zhan F, Ma X, Wang D, Xu W, Wu G, Gao GF, Tan W; China Novel Coronavirus Investigating and Research Team. A Novel Coronavirus from Patients with Pneumonia in China, 2019. N Engl J Med. 2020 Feb 20;382(8):727-733. doi: 10.1056/NEJMoa2001017. Epub 2020 Jan 24. PMID 31978945
- [Background] Wu F, Zhao S, Yu B, Chen YM, Wang W, Song ZG, Hu Y, Tao ZW, Tian JH, Pei YY, Yuan ML, Zhang YL, Dai FH, Liu Y, Wang QM, Zheng JJ, Xu L, Holmes EC, Zhang YZ. A new coronavirus associated with human respiratory disease in China. Nature. 2020 Mar;579(7798):265-269. doi: 10.1038/s41586-020-2008-3. Epub 2020 Feb 3. PMID 32015508
- [Background] Wu F, Zhao S, Yu B, Chen YM, Wang W, Song ZG, Hu Y, Tao ZW, Tian JH, Pei YY, Yuan ML, Zhang YL, Dai FH, Liu Y, Wang QM, Zheng JJ, Xu L, Holmes EC, Zhang YZ. Author Correction: A new coronavirus associated with human respiratory disease in China. Nature. 2020 Apr;580(7803):E7. doi: 10.1038/s41586-020-2202-3. PMID 32296181
- [Background] Young BE, Ong SWX, Kalimuddin S, Low JG, Tan SY, Loh J, Ng OT, Marimuthu K, Ang LW, Mak TM, Lau SK, Anderson DE, Chan KS, Tan TY, Ng TY, Cui L, Said Z, Kurupatham L, Chen MI, Chan M, Vasoo S, Wang LF, Tan BH, Lin RTP, Lee VJM, Leo YS, Lye DC; Singapore 2019 Novel Coronavirus Outbreak Research Team. Epidemiologic Features and Clinical Course of Patients Infected With SARS-CoV-2 in Singapore. JAMA. 2020 Apr 21;323(15):1488-1494. doi: 10.1001/jama.2020.3204. PMID 32125362
- [Background] Spiteri G, Fielding J, Diercke M, Campese C, Enouf V, Gaymard A, Bella A, Sognamiglio P, Sierra Moros MJ, Riutort AN, Demina YV, Mahieu R, Broas M, Bengner M, Buda S, Schilling J, Filleul L, Lepoutre A, Saura C, Mailles A, Levy-Bruhl D, Coignard B, Bernard-Stoecklin S, Behillil S, van der Werf S, Valette M, Lina B, Riccardo F, Nicastri E, Casas I, Larrauri A, Salom Castell M, Pozo F, Maksyutov RA, Martin C, Van Ranst M, Bossuyt N, Siira L, Sane J, Tegmark-Wisell K, Palmerus M, Broberg EK, Beaute J, Jorgensen P, Bundle N, Pereyaslov D, Adlhoch C, Pukkila J, Pebody R, Olsen S, Ciancio BC. First cases of coronavirus disease 2019 (COVID-19) in the WHO European Region, 24 January to 21 February 2020. Euro Surveill. 2020 Mar;25(9):2000178. doi: 10.2807/1560-7917.ES.2020.25.9.2000178. PMID 32156327
- [Background] Mousavi SH, Shah J, Giang HTN, Al-Ahdal TMA, Zahid SU, Temory F, Paikan FM, Karimzadeh S, Huy NT. The first COVID-19 case in Afghanistan acquired from Iran. Lancet Infect Dis. 2020 Jun;20(6):657-658. doi: 10.1016/S1473-3099(20)30231-0. Epub 2020 Mar 23. No abstract available. PMID 32213330
- [Background] Silverstein WK, Stroud L, Cleghorn GE, Leis JA. First imported case of 2019 novel coronavirus in Canada, presenting as mild pneumonia. Lancet. 2020 Feb 29;395(10225):734. doi: 10.1016/S0140-6736(20)30370-6. Epub 2020 Feb 13. No abstract available. PMID 32061312
- [Background] Holshue ML, DeBolt C, Lindquist S, Lofy KH, Wiesman J, Bruce H, Spitters C, Ericson K, Wilkerson S, Tural A, Diaz G, Cohn A, Fox L, Patel A, Gerber SI, Kim L, Tong S, Lu X, Lindstrom S, Pallansch MA, Weldon WC, Biggs HM, Uyeki TM, Pillai SK; Washington State 2019-nCoV Case Investigation Team. First Case of 2019 Novel Coronavirus in the United States. N Engl J Med. 2020 Mar 5;382(10):929-936. doi: 10.1056/NEJMoa2001191. Epub 2020 Jan 31. PMID 32004427
- [Background] Kim JY, Choe PG, Oh Y, Oh KJ, Kim J, Park SJ, Park JH, Na HK, Oh MD. The First Case of 2019 Novel Coronavirus Pneumonia Imported into Korea from Wuhan, China: Implication for Infection Prevention and Control Measures. J Korean Med Sci. 2020 Feb 10;35(5):e61. doi: 10.3346/jkms.2020.35.e61. PMID 32030925
- [Background] Ghinai I, McPherson TD, Hunter JC, Kirking HL, Christiansen D, Joshi K, Rubin R, Morales-Estrada S, Black SR, Pacilli M, Fricchione MJ, Chugh RK, Walblay KA, Ahmed NS, Stoecker WC, Hasan NF, Burdsall DP, Reese HE, Wallace M, Wang C, Moeller D, Korpics J, Novosad SA, Benowitz I, Jacobs MW, Dasari VS, Patel MT, Kauerauf J, Charles EM, Ezike NO, Chu V, Midgley CM, Rolfes MA, Gerber SI, Lu X, Lindstrom S, Verani JR, Layden JE; Illinois COVID-19 Investigation Team. First known person-to-person transmission of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in the USA. Lancet. 2020 Apr 4;395(10230):1137-1144. doi: 10.1016/S0140-6736(20)30607-3. Epub 2020 Mar 13. PMID 32178768
- [Background] Wiersinga WJ, Rhodes A, Cheng AC, Peacock SJ, Prescott HC. Pathophysiology, Transmission, Diagnosis, and Treatment of Coronavirus Disease 2019 (COVID-19): A Review. JAMA. 2020 Aug 25;324(8):782-793. doi: 10.1001/jama.2020.12839. PMID 32648899
- [Result] Organizational impact of an ID NOW™ COVID-19 point-of-care testing for SARS-CoV2 detection in a maternity ward Jean-Claude Nguyen Van, Benoît Pilmis, Amir Khaterchi, Olivier Billuart, Gauthier Péan De Ponfilly, Alban Le Monnier, Elie Azria, Assaf Mizrahi
- See also: https://splf.fr/wp-content/uploads/2020/04/Societe-franc%CC%A7aise-de-microbiologie-Recommandations-pour-le-diagnostic-specifique-du-COVID-1-en-biologie-delocalisee-Version-1-09-04-20.pdf — https://splf.fr/wp-content/uploads/2020/04/Societe-franc%CC%A7aise-de-microbiologie-Recommandations-pour-le-diagnostic-specifique-du-COVID-1-en-biologie-delocalisee-Version-1-09-04-20.pdf
- See also: https://www.medrxiv.org/content/10.1101/2022.08.29.22279161v1.full.pdf — https://www.medrxiv.org/content/10.1101/2022.08.29.22279161v1.full.pdf